CLINICAL TRIAL: NCT04092582
Title: A Phase IIa, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of MTPS9579A in Patients With Asthma Requiring Inhaled Corticosteroids and a Second Controller
Brief Title: A Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of MTPS9579A in Patients With Asthma Requiring Inhaled Corticosteroids and a Second Controller
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GB41149; 2019-000795-41 (EudraCT Number)
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTPS9579A (Experimental)
  Interventions: Drug: MTPS9579A
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MTPS9579A — MTPS9579A IV infusion will be administered at the randomization visit (Week 2), Week 6, and every 4 weeks through Week 46.
  Arms: MTPS9579A
Drug: Placebo — Placebo matching MTPS9579A will be administered at the randomization visit (Week 2), Week 6, and every 4 weeks thereafter through Week 46.
  Arms: Placebo

SUMMARY:
This is a Phase IIa, randomized, placebo-controlled, double-blind, multicenter, two-arm study to evaluate the efficacy, safety, and pharmacokinetics of MTPS9579A as an add-on therapy in patients with uncontrolled moderate to severe asthma who are receiving daily ICS therapy and at least one of the following additional controller medications: long-acting beta-agonist (LABA), leukotriene modulator (leukotriene modifier [LTM] or leukotriene receptor antagonist [LTRA]), long-acting muscarinic antagonist (LAMA), or long-acting theophylline preparation.

ELIGIBILITY:
Inclusion Criteria:

* Documented physician-diagnosed asthma for at least 12 months prior to screening
* Treatment with asthma controller therapy (daily ICS [fluticasone propionate or equivalent] and at least one additional controller therapy [LABA, LAMA, LTM/LTRA]) for >= 3 months prior to screening, with no changes within 4 weeks prior to screening or during the screening period and no anticipated changes in controller dosing regimens throughout the study
* Documented history of >= 2 asthma exacerbation within the 12 months prior to screening while on daily ICS maintenance therapy
* For women of childbearing potential: agreement to remain abstinent or use contraception For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm

Exclusion Criteria:

* History or evidence of vocal cord dysfunction, reactive airways dysfunction syndrome, hyperventilation associated with panic attacks, or other mimics of asthma
* History or evidence of significant respiratory disease other than asthma, including occupational asthma, aspirin-sensitive asthma, asthma-chronic obstructive pulmonary disease (COPD) overlap syndrome, bronchiolitis, interstitial lung disease, or COPD
* Current smoker, electronic cigarette (e-cigarette) user, former smoker with smoking history of > 10 pack-years, former e-cigarette user with an e-cigarette history of at least daily use for >=10 years, or unwilling to abstain from smoking and/or e-cigarette use from the time of consent through the completion of the study
* History or evidence of any clinically significant medical condition/disease or abnormalities in laboratory tests that, in the investigator's judgment, precludes the patient's safe participation and completion of the study, or interferes with the conduct and interpretation of the study
* Active malignancy or history of malignancy within 5 years of screening, except for appropriately treated non-melanoma skin carcinoma, cervical carcinoma in situ, breast ductal carcinoma in situ, or Stage I uterine cancer
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 60 days after the final dose of MTPS9579A
* Positive for TB at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (27):
- United States (8):
  - Kern Research, Bakersfield, California
  - Allergy & Asthma Medical Group of the Bay Area, Walnut Creek, California
  - Florida Ctr-Allergy & Asthma, Miami, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - Toledo Inst of Clin Research, Toledo, Ohio
  - OK Clinical Research, Edmond, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
- Argentina (4):
  - Fundacion Cidea, Buenos Aires
  - Centro Médico Dra. Cristina de Salvo, Buenos Aires
  - CARE - Centro de Alergia y Enfermedades Respiratorias, CABA
  - Centro Respiratorio Quilmes, Quilmes
- Germany (5):
  - Research Center for Medical Studies RCMS, Berlin
  - IKF Pneumologie, Frankfurt am Main
  - Pneumologicum, Hanover
  - BAG Prof Dr G Hoheisel Dr A Bonitz, Leipzig
  - SMO.MD GmbH, Zentrum für klinische Studien, Magdeburg
- Peru (2):
  - Clinica Providencia (Inverconsult Sociedad Anonima), Lima
  - Clinica Ricardo Palma; THORAX, Lima
- Poland (8):
  - Centrum Medycyny Oddechowej Robert M. Mróz, Bialystok
  - Centrum Medyczne ALL-MED, Krakow
  - Malopolskie Centrum Alergologii, Krakow
  - SPZOZ Uniwersytecki Szpital Kliniczny nr 1 im. Norberta Barlickiego Uniwersytetu Medycznego w Lodzi, Lodz
  - Ostrowieckie Centrum Medyczne Spolka Cywilna Anna Olec-Cudzik; Krzysztof Cudzik, Ostrowiec Swietokrzysk
  - Centrum Alergologii Teresa Hofman, Poznan
  - PULMAG Grzegorz Gasior Marzena Kociolek Spolka Cywilna, Sosnowiec
  - ALL-MED Specjalistyczna Opieka Medyczna, Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study-Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 26 investigative sites in 5 countries (Argentina, Germany, Peru, Poland, and the United States) from 31 October 2019 to 19 May 2022.
Pre-assignment Details: This study included a 2-week single-blind placebo run-in period. A total of 135 participants were randomized in double-blind treatment period. Of the 135 participants randomized, 134 participants received at least one dose of study drug and their intended treatment.
Groups:
- MTPS9579A, 1800 mg: Participants with uncontrolled moderate to severe asthma received Placebo, given as intravenous (IV) infusion, for 14 days in the Placebo run-in period. Participants then received MTPS9579A, 1800 mg, given as IV infusion at randomization (Week 2), Week 6, and every 4 weeks thereafter through Week 46.
- Placebo: Participants with uncontrolled moderate to severe asthma received Placebo, given as IV infusion, for 14 days in the Placebo run-in period. Participants received MTPS9579A matching placebo, given as IV infusion at randomization (Week 2), Week 6, and every 4 weeks thereafter through Week 46.
Period: Overall Study
Arm/Group | MTPS9579A, 1800 mg | Placebo
Started | 69 | 66
Safety Population (The safety analysis population included all randomized participants who received at least one dose of study drug during the 48-week double-blind treatment period.) | 69 | 65
Completed | 64 | 63
Not Completed | 5 | 3
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Enrolled but Failed to Meet Randomization Criteria; Excluded from Study Analysis | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat population (mITT) population included all randomized participants who received at least one dose of study treatment.
Groups:
- MTPS9579A, 1800 mg: Participants with uncontrolled moderate to severe asthma received Placebo, given as IV infusion, for 14 days in the Placebo run-in period. Participants then received MTPS9579A,1800 mg, given as IV infusion at randomization (Week 2), Week 6, and every 4 weeks thereafter through Week 46.
- Total: Total of all reporting groups
Arm/Group | MTPS9579A, 1800 mg | Placebo | Total
Number analyzed (Participants) | 69 | 65 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (12.0) | 52.9 (13.2) | 53.8 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 34 | 73
  Male | 30 | 31 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 22
  Not Hispanic or Latino | 59 | 53 | 112
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 62 | 59 | 121
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to First Composite Asthma Exacerbations (CompEX) Event
Description: CompEX is defined as time from randomization to first asthma exacerbation or diary worsening during the treatment period.
  Asthma exacerbation was defined as new or increased asthma symptoms (wheezing, coughing, dyspnea, chest tightness, and/or nighttime awakenings due to these symptoms) that resulted in one or both of the following: Hospitalization or emergency department visit with administration of systemic corticosteroid treatment; Treatment with systemic corticosteroids for at least 3 days, or a long-acting depot corticosteroid preparation with a therapeutic effectiveness of at least 3 days. Diary worsening is based on the occurrence of prespecified changes in the following six parameters: morning peak expiratory flow rate (PEFR), evening PEFR, morning symptom score, evening symptom score, morning short-acting rescue therapy use, and evening short-acting rescue therapy use. Hazard ratio was used for the analysis.
Time Frame: Randomization [Week 2] to end of treatment (EOT) [Week 50]
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- MTPS9579A, 1800 mg: Participants with uncontrolled moderate to severe asthma received Placebo, given as IV infusion, for 14 days in the Placebo run-in period. Participants then received MTPS9579A, 1800 mg, given as IV infusion at randomization (Week 2), Week 6, and every 4 weeks thereafter through Week 46.
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 69 | 65
weeks | NA [31.3 to NA] — The data for median upper limit of confidence interval (CI) was not estimable due to insufficient number of participants with events. | 45.4 [19.0 to NA] — The data for upper limit of CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: MTPS9579A, 1800 mg vs Placebo; Test type: Superiority; p = 0.6835, Regression, Cox; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.55 to 1.47]

2. Secondary Outcome: Rate of Asthma Exacerbations
Description: The number of asthma exacerbations per year was reported for this outcome measure. Asthma exacerbation was defined as new or increased asthma symptoms (wheezing, coughing, dyspnea, chest tightness, and/or nighttime awakenings due to these symptoms) that resulted in one or both of the following: Hospitalization or emergency department visit with administration of systemic corticosteroid treatment; Treatment with systemic corticosteroids for at least 3 days, or a long-acting depot corticosteroid preparation with a therapeutic effectiveness of at least 3 days. Poisson regression was used for the analysis.
Time Frame: Randomization [Week 2] to Week 50
Population: mITT population included all randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Asthma exacerbations per patient-year
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 69 | 65
Asthma exacerbations per patient-year | 0.4689 | 0.4267
Statistical Analysis 1: Comparison: MTPS9579A, 1800 mg vs Placebo; Test type: Superiority; p = 0.7648, Poisson regression; Rate Ratio = 1.0989, 95% CI 2-sided [0.5925 to 2.0381]

3. Secondary Outcome: Time to First Asthma Exacerbation
Description: The time from randomization to first asthma exacerbation was measured. Asthma exacerbation was defined as new or increased asthma symptoms (wheezing, coughing, dyspnea, chest tightness, and/or nighttime awakenings due to these symptoms) that resulted in one or both of the following: Hospitalization or emergency department visit with administration of systemic corticosteroid treatment; Treatment with systemic corticosteroids for at least 3 days, or a long-acting depot corticosteroid preparation with a therapeutic effectiveness of at least 3 days. Cox regression was used for the analysis.
Time Frame: Randomization [Week 2] to Week 50
Population: mITT population included all randomized participants who received at least one dose of study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 69 | 65
weeks | NA [NA to NA] — The data for median, lower and upper limit of CI was not estimable due to insufficient number of participants with events. | NA [NA to NA] — The data for median, lower and upper limit of CI was not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: MTPS9579A, 1800 mg vs Placebo; Test type: Superiority; p = 0.5248, Regression, Cox; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.43 to 1.54]

4. Secondary Outcome: Absolute Change From Randomization in Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1) at Week 50
Description: FEV1 is calculated as the volume of air forcibly exhaled in one second as measured by a spirometer. Estimates are based on a mixed model for repeated measures (MMRM) analysis with an unstructured covariance matrix. The model used the absolute change pre-bronchodilator FEV1 as the response variable and included terms for treatment arm, study visit, treatment arm by study visit interaction, baseline FEV1 as well as its interaction with study visit, in addition to the stratification factors: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/microliter (uL)), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region.
Time Frame: Randomization [Week 2] to Week 50
Population: mITT population included all randomized participants who received at least one dose of study treatment. Overall number of participants analyzed are the number of participants available for analysis.
Measure: Mean (Standard Error); unit: liters
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 62 | 61
liters | 0.11 (0.034) | 0.03 (0.034)
Statistical Analysis 1: Comparison: MTPS9579A, 1800 mg vs Placebo; Test type: Superiority; p = 0.1250, Mixed model for repeated measures (MMRM)

5. Secondary Outcome: Relative Percent Change From Randomization in Pre-Bronchodilator FEV1 at Week 50
Description: FEV1 was the volume of air exhaled in the first second of a forced exhalation as measured by spirometer. Measurements were performed before use of bronchodilator. Estimates are based on a mixed model for repeated measures (MMRM) analysis with an unstructured covariance matrix. The model used the relative change pre-bronchodilator FEV1 as the response variable and included terms for treatment arm, study visit, treatment arm by study visit interaction, baseline FEV1 as well as its interaction with study visit, in addition to the stratification factors: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region. Relative change (%) in FEV1 = (absolute change in FEV1 / baseline FEV1) x 100.
Time Frame: Randomization [Week 2] to Week 50
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 62 | 61
percent change | 6.44 (1.894) | 3.15 (1.921)
Statistical Analysis 1: Comparison: MTPS9579A, 1800 mg vs Placebo; Test type: Superiority; p = 0.2249, Mixed model for repeated measures (MMRM)

6. Secondary Outcome: Absolute Change From Randomization in Fractional Exhaled Nitric Oxide (FeNO) at Week 50
Description: FeNO is a volatile marker of airway inflammation that decreases with inhaled corticosteroid treatment. The measurements recorded were according to standardized procedures by the American Thoracic Society. Estimates are based on a mixed model for repeated measures (MMRM) analysis with an unstructured covariance matrix. The model used the absolute change pre-bronchodilator FeNO as the response variable and included terms for treatment arm, study visit, treatment arm by study visit interaction, baseline FeNO as well as its interaction with study visit, in addition to the stratification factors: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region.
Time Frame: Randomization [Week 2] to Week 50
Population: as for outcome 4
Measure: Mean (Standard Error); unit: parts per billion (ppb)
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 57 | 54
parts per billion (ppb) | -1.67 (2.722) | -1.52 (2.791)
Statistical Analysis 1: Comparison: MTPS9579A, 1800 mg vs Placebo; Test type: Superiority; p = 0.9693, Mixed model for repeated measures (MMRM)

7. Secondary Outcome: Relative Percent Change From Randomization in FeNO at Week 50
Description: FeNO is a volatile marker of airway inflammation that decreases with inhaled corticosteroid treatment. The measurements recorded were according to standardized procedures by the American Thoracic Society. Relative change (%) in FeNO = (absolute change in FeNO / baseline FeNO) x 100. Estimates are based on a mixed model for repeated measures (MMRM) analysis with an unstructured covariance matrix. The model used the absolute change pre-bronchodilator FeNO as the response variable and included terms for treatment arm, study visit, treatment arm by study visit interaction, baseline FeNO as well as its interaction with study visit, in addition to the stratification factors: blood eosinophil level at visit 1 (<150, >=150 to <=300, >300 cells/uL), number of asthma exacerbations requiring the use of systemic corticosteroids within the 12 months prior to the study entry (1 or >=2 events), and geographic region.
Time Frame: Randomization [Week 2] to Week 50
Population: as for outcome 4
Measure: Mean (Standard Error); unit: percent change
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 57 | 54
percent change | 26.02 (10.223) | 26.29 (10.482)
Statistical Analysis 1: Comparison: MTPS9579A, 1800 mg vs Placebo; Test type: Superiority; p = 0.9855, Mixed model for repeated measures (MMRM)

8. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product.
Time Frame: Up to approximately Week 58
Population: The safety analysis population included all randomized participants who received at least one dose of study drug during the 48-week double-blind treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 69 | 65
percentage of participants | 79.7 | 86.2

9. Secondary Outcome: Area Under Concentration-Time Curve for the First Dosing Interval (AUClast) of MTPS9579A
Time Frame: Randomization [Week 2] to Week 6
Population: PK-evaluable population includes all participants who had at least one evaluable PK sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*ug/mL
Arm/Group | MTPS9579A, 1800 mg
Number analyzed (Participants) | 69
day*ug/mL | 5263.14 (83.6)

10. Secondary Outcome: Maximum Serum Concentration (Cmax) for the First Dosing Interval of MTPS9579A
Time Frame: 2-hour post-dose on Week 2
Population: PK-evaluable population includes all participants who had at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | MTPS9579A, 1800 mg
Number analyzed (Participants) | 69
ug/mL | 419 (51.4)

11. Secondary Outcome: Steady State Cmax of MTPS9579A
Time Frame: 2-hour post-dose on Week 14
Population: PK-evaluable population includes all participants who had at least one evaluable PK sample
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | MTPS9579A, 1800 mg
Number analyzed (Participants) | 69
ug/mL | 735 (31.0)

12. Secondary Outcome: Maximum Time to Serum Concentration (Tmax) of MTPS9579A
Time Frame: Pre-dose and 2-hour post-dose on Week 2
Population: PK-evaluable population includes all participants who had at least one evaluable PK sample.
Measure: Median (Standard Deviation); unit: day
Arm/Group | MTPS9579A, 1800 mg
Number analyzed (Participants) | 69
day | 0.12 (3.41)

13. Secondary Outcome: Trough Serum Concentration (Ctrough) Accumulation Ratio of MTPS9579A
Description: The accumulation ratio is calculated by taking the individual ratio of the Ctrough at Week 14 to the Ctrough at Week 6.
Time Frame: Predose on Weeks 6 and 14
Population: PK-evaluable population includes all participants who had at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | MTPS9579A, 1800 mg
Number analyzed (Participants) | 69
ratio | 1.93 (28.3)

14. Secondary Outcome: Steady State Ctrough of MTPS9579A
Time Frame: Pre-dose on Week 14
Population: PK-evaluable population includes all participants who had at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | MTPS9579A, 1800 mg
Number analyzed (Participants) | 69
ug/mL | 226 (45.4)

15. Secondary Outcome: Percentage of Participants With Anti-Drug Antibodies (ADA) to MTPS9579A
Description: Treatment Emergent ADA is (a) negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result, OR (b) positive ADA result at baseline and one or more post-baseline titer results that are at least 0.60 titer unit (t.u.) greater than the baseline titer result.
Time Frame: Pre-dose Week 54
Population: The immunogenicity analysis population included all participants with at least one ADA assessment.
Measure: Number; unit: percentage of participants
Arm/Group | MTPS9579A, 1800 mg | Placebo
Number analyzed (Participants) | 68 | 65
percentage of participants | 5.9 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately Week 58
Description: All cause mortality data was collected for all enrolled participants and serious adverse events (SAE) and other adverse events (AE) was collected for Safety analysis population. The safety analysis population included all randomized participants who received at least one dose of study drug during the 48-week double-blind treatment period.
Arm/Group | MTPS9579A, 1800 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 1/69 | 1/66
Serious Adverse Events (participants affected / at risk) | 5/69 | 4/65
Other Adverse Events (participants affected / at risk) | 32/69 | 38/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTPS9579A, 1800 mg (N=69) | Placebo (N=65)
Accidental death (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTPS9579A, 1800 mg (N=69) | Placebo (N=65)
COVID-19 (Infections and infestations) | 6 (6) | 6 (6)
Nasopharyngitis (Infections and infestations) | 4 (5) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 5 (6) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 (31) | 24 (33)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)

LIMITATIONS AND CAVEATS:
Enrollment was halted on 08 April 2020 in response to the emerging pandemic and concerns regarding data integrity (e.g., missed study doses and visits). The trial was restarted on 22 June 2020.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-09-18): https://cdn.clinicaltrials.gov/large-docs/82/NCT04092582/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-30): https://cdn.clinicaltrials.gov/large-docs/82/NCT04092582/SAP_001.pdf